CLINICAL TRIAL: NCT01514136
Title: CP216: An Exploratory Investigation of Convex Ostomy Devices
Brief Title: An Investigation of Ostomy Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CP216
Record Dates: First submitted 2012-01-10; First posted 2012-01-20 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One arm (Experimental): The arm consists of two periods: in period one, products are tested in the order A, B, C, D, and in period two, products are tested in the order A*, B*, C*, D*.
  Interventions: Device: Ostomy appliance: convex 1-piece drainable

INTERVENTIONS:
Device: Ostomy appliance: convex 1-piece drainable — 8 variations of an ostomy devices are tested

SUMMARY:
Coloplast A/S has developed a new ostomy device in 8 versions.

The primary objective of this investigation is to assess and compare the degree of leakage when using the 8 different devices.

The secondary objective is to investigate several performance and safety parameters of the various devices.

The aim of the primary and secondary objectives is to acquire more knowledge about the performance of the newly developed device and inspiration for their further development, if needed.

Given that the investigation is exploratory, pass/fail criteria are not relevant. The investigation result will provide knowledge useful for continued decision-making/device development.

The investigation is designed as a non-blinded, controlled, exploratory investigation that includes a total of 30-40 Danish ileostomy users.

Each subject will test a maximum of 4 convex devices in two rounds of each 4 weeks. Each device will be tested for 7 (± 2) days.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have signed the declaration of informed consent
* Have an ileostomy in a concave area
* Have had an ileostomy for at least three months
* Have used convex plates (for convex users) or flat plates (for flat plate users) for the last month
* Be users of 1-piece or 2-piece open ostomy devices
* Have an ileostomy with a diameter of less than 33 mm

Exclusion Criteria:

* Are pregnant or breast-feeding
* Have a double-loop ileostomy
* Have known hypersensitivity or allergy to the devices' component ingredients
* Are receiving/have received radiation treatment and/or chemotherapy within the last 3 months.
* Are receiving/have received local peristomal or systemic steroid treatment within the last month
* Suffer from peristomal skin problems that preclude participation in the investigation (assessed by the investigation nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject were recruited through the Coloplast A/S user database in Denmark.
Pre-assignment Details: The investigation consisted of two periods: in the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts, Test A*-D*, were developed and tested. The test products were not randomised. The test order in first round was Test A - Test D and in second round it was Test A*-Test D*.
Groups:
- Test A: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test A was a newly developed concept by Coloplast A/S for the first round.
- Test B: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test B was a newly developed concept by Coloplast A/S for the first round.
- Test C: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test C was a newly developed concept by Coloplast A/S for the first round.
- Test D: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test D was a newly developed concept by Coloplast A/S for the first round.
- Test A*: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test A* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test B*: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test B* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test C*: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test C* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test D*: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Therefore the participant flow is divided by the test products and not for each period.
  Test D* was a newly developed optimized concept by Coloplast A/S for the second round.
Period: Test Period 1; Test A
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 25 (26 subjects tested Test A) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Break from study holiday | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 1; Test B
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 24 (2 new subjects were entered the investigation) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 1; Test C
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 0 | 24 (1 new subject was included in the investigation) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 24 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 1; Test D
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 0 | 0 | 26 (The two subject that were on holiday after test A re-entered the investigation) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Subject took a break due to holiday | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Test Period 2; Test A*
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 0 | 0 | 0 | 28 (4 new subjects were included in the investigation) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 26 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Holiday | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Test Period 2; Test B*
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 0 | 0 | 0 | 0 | 28 (Two subjects did not test test A*, but had a break and continued again on Test B*) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Test Period 2; Test C*
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — holiday | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Test Period; Test D*
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Convex Product Users: Subjects who usually use a convex product
- Flat Product Users: Subjects who usually use a flat product
- Total: Total of all reporting groups
Arm/Group | Convex Product Users | Flat Product Users | Total
Number analyzed (Participants) | 23 | 9 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.9) | 64.4 (7.5) | 60.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 5 | 23
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage under the baseplate was measured on a 24-point scale where 0 point was the best possible outcome with no leakage under the baseplate and 24-point was the worst possible outcome with leakage under the whole plate.
  The scale was developed by Coloplast A/S
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Test A - Convex Product Users; Test A - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test A was a newly developed concept by Coloplast A/S for the first round.
- Test B - Convex Product Users; Test B - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test B was a newly developed concept by Coloplast A/S for the first round.
- Test C - Convex Product Users; Test C - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test C was a newly developed concept by Coloplast A/S for the first round.
- Test D - Convex Product Users; Test D - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test D was a newly developed concept by Coloplast A/S for the first round.
- Test A* - Convex Product Users; Test A* - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test A* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test B* - Convex Product Users; Test B* - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test B* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test C* - Convex Product Users; Test C* - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test C* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test D* - Convex Product Users; Test D* - Flat Product Users: The investigation was set up with two different periods. In the first period the newly developed concepts, Test A-D, were tested. Based on the results, four new concepts were developed and tested, Test A* - D*.
  Two subject populations were included in the investigation: subjects using flat ostomy products and subjects using convex ostomy products.
  Test D* was a newly developed optimized concept by Coloplast A/S for the second round.
Arm/Group | Test A - Convex Product Users | Test B - Convex Product Users | Test C - Convex Product Users | Test D - Convex Product Users | Test A* - Convex Product Users | Test B* - Convex Product Users | Test C* - Convex Product Users | Test D* - Convex Product Users | Test A - Flat Product Users | Test B - Flat Product Users | Test C - Flat Product Users | Test D - Flat Product Users | Test A* - Flat Product Users | Test B* - Flat Product Users | Test C* - Flat Product Users | Test D* - Flat Product Users
Number analyzed (Participants) | 18 | 19 | 19 | 19 | 19 | 20 | 18 | 16 | 7 | 5 | 5 | 7 | 9 | 8 | 8 | 7
Number analyzed (baseplates) | 99 | 98 | 111 | 92 | 104 | 89 | 87 | 86 | 36 | 32 | 31 | 43 | 43 | 42 | 41 | 35
units on a scale | 4.2 (0.6) | 4.3 (0.8) | 4.4 (0.7) | 4.3 (0.8) | 3.4 (0.7) | 2.9 (0.6) | 3.3 (0.7) | 4.1 (0.8) | 2.1 (1.4) | 0.1 (0.04) | 0.1 (0.1) | 2.4 (1.3) | 3.1 (1.5) | 3.6 (1.8) | 3.8 (1.8) | 3.0 (1.6)

ADVERSE EVENTS:
Groups:
- Test A: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test A was a newly developed concept by Coloplast A/S for the first round.
- Test B: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test B was a newly developed concept by Coloplast A/S for the first round.
- Test C: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test C was a newly developed concept by Coloplast A/S for the first round.
- Test D: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test D was a newly developed concept by Coloplast A/S for the first round.
- Test A*: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test A* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test B*: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test B* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test C*: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test C* was a newly developed optimized concept by Coloplast A/S for the second round.
- Test D*: The investigation was set up with two different periods. In the first period the newly developed concepts Test A-D were tested based on the results four new products were developed and tested concept Test A* - D*.
  Test D* was a newly developed optimized concept by Coloplast A/S for the second round.
Arm/Group | Test A | Test B | Test C | Test D | Test A* | Test B* | Test C* | Test D*
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/24 | 0/26 | 1/28 | 0/28 | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 8/26 | 6/24 | 4/24 | 3/26 | 3/28 | 3/28 | 1/26 | 3/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A (N=26) | Test B (N=24) | Test C (N=24) | Test D (N=26) | Test A* (N=28) | Test B* (N=28) | Test C* (N=26) | Test D* (N=23)
Chemotherapy, cancer in lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to the product
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A (N=26) | Test B (N=24) | Test C (N=24) | Test D (N=26) | Test A* (N=28) | Test B* (N=28) | Test C* (N=26) | Test D* (N=23)
Perstomal skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) — Related to the product
Cold or influenza (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Not related to the product
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to the product
Protocol deviation/not defined (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Related or possibly related to the product
Cancer, therapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to the product
Infection, tooth (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to the product
Liver values, increased (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to the product

LIMITATIONS AND CAVEATS:
This was an exploratory investigation where the participating subjects had to test 8 different test products. A small number of subjects were analysed from two different populations (convex product/flat product users).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes